CLINICAL TRIAL: NCT03730610
Title: Modelling Systemic Cross-talk Between Brain, Gut, and Peripheral Tissues in Glucose Homeostasis: Exercise Training and Public Health
Brief Title: Systemic Cross-talk Between Brain, Gut, and Peripheral Tissues in Glucose Homeostasis: Effects of Exercise Training
Acronym: CROSSYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of Helsinki (Other); University of Eastern Finland (Other); Turku University Hospital (Other Government); Academy of Finland (Other); Finnish Cultural Foundation (Other); Diabetes Research Foundation, Finland (Other); Juho Vainio Foundation (Other)
Responsible Party: Principal Investigator, Jarna Hannukainen, Adjunct Professor, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 317332
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Insulin Resistance; Type2 Diabetes; Exercise Training
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise Training for six months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Experimental): Six months of exercise training
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Subjects are required to exercise four times a week during six months. Exercise training consists of endurance training, resistance training and high-intensity interval training adjusted to subject's fitness level.

SUMMARY:
Obesity and insulin resistance are worldwide epidemic and taking a major public health toll. Obesity also increases the risk for cognitive impairment which is also an increasing medical, societal, and economic challenge. The ultimate goal of this proposal is to develop a statistical model to assess systemic cross-talk between brain, peripheral tissues, gut microbiota and glucose metabolism. Integrated with exercise training intervention the results will be utilized to provide disease risk profiling and personalized predictions of exercise training as a drug free treatment for insulin resistance and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* monozygotic twins
* body mass index (BMI) difference ≥ 2 kg/m2 and/or type 2 diabetes
* At least one co-twin is overweight (BMI > 25 kg/m2)

Exclusion Criteria:

* BMI > 60 kg/m2
* body weight > 170 kg
* waist circumference > 150 cm
* mental disorder or poor compliance
* eating disorder or excessive use of alcohol
* active ulcus disease
* diabetes requiring insulin treatment or fasting glucose > 10 mmol/l
* pregnancy
* past dose of radiation
* claustrophobia
* presence of ferromagnetic objects that would make MRI contraindicated

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Effects of exercise training - brain glucose uptake | The change from baseline to 6 months
  Brain glucose uptake (micromol/100g/min) is measured with positron emission tomography (PET) with [18F]-labelled fluoro-deoxy-glucose (FDG) tracer.
Effects of exercise training - brain inflammation | The change from baseline to 6 months
  Brain inflammation (dimensionless; standistibution volume ratio) is measured with positron emission tomography (PET) with PK11195 tracer

SECONDARY OUTCOMES:
Effects of exercise training - liver glucose uptake | The change from baseline to 6 months
  Liver glucose uptake (micromol/100g/min) is measured with positron emission tomography (PET) with [18F]-labelled fluoro-deoxy-glucose (FDG) tracer
Effects of exercise training - adipose tissue glucose uptake | The change from baseline to 6 months
  Adipose tissue glucose uptake (micromol/100g/min) is measured with positron emission tomography (PET) with [18F]-labelled fluoro-deoxy-glucose (FDG) tracer
Effects of exercise training - whole-body insulin sensitivity | The change from baseline to 6 months
  Whole-body insulin sensitivity (M-value; micromol/100g/min) during the hyperinsulinemic euglycemic clamp
Effects of exercise training - ectopic fat | The change from baseline to 6 months
  Ectopic fat content (%) is measured using magnetic resonance spectroscopy (MRS)

CONTACTS AND LOCATIONS:
Overall Officials: Jarna Hannukainen, PhD, Principal Investigator — Turku PET Cente, University of Turku, Finland
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided
IPD of the main outcome measures will be opened if possible to such as extent that individuals cannot be identified.

REFERENCES:
- [Derived] Heiskanen MA, Honkala SM, Hentila J, Ojala R, Lautamaki R, Koskensalo K, Lietzen MS, Saunavaara V, Saunavaara J, Helmio M, Loyttyniemi E, Nummenmaa L, Collado MC, Malm T, Lahti L, Pietilainen KH, Kaprio J, Rinne JO, Hannukainen JC. Systemic cross-talk between brain, gut, and peripheral tissues in glucose homeostasis: effects of exercise training (CROSSYS). Exercise training intervention in monozygotic twins discordant for body weight. BMC Sports Sci Med Rehabil. 2021 Feb 24;13(1):16. doi: 10.1186/s13102-021-00241-z. PMID 33627179